CLINICAL TRIAL: NCT00896259
Title: Effects of a Late Phase Education and Exercise Program Following Total Hip Arthroplasty: A Pilot Project
Brief Title: Effects of a Late Phase Exercise Program Following Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Canadian Orthopaedic Foundation (Other)
Responsible Party: Principal Investigator, Kim Parker, Rehabilitation Engineer, Nova Scotia Health Authority
Other Study IDs: CDHA-RS/2007-057
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Total Hip Arthroplasty
Keywords: Unilateral total hip arthroplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- THA control: those with THA not participating in exercise and education program
- THA exercise: those with THA and participating in exercise and education program
  Interventions: Other: home based exercise and education program
- healthy control: Healthy control, people with no lower limb gait abnormalities

INTERVENTIONS:
Other: home based exercise and education program — Individual assessment with physiotherapist with educational information, exercise instruction and prescription provided. Instructed to perform home exercises and walking for 12 weeks. Will be individually tailored to participants, bi-monthly phone calls will be used to monitor and facilitate exercise and walking progression .
  Groups: THA exercise

SUMMARY:
A group of orthopedic physiotherapists have developed a late phase program to educate and instruct total hip replacement patients in progressive exercises appropriate for their level of recovery. The components of this program include an educational presentation, individual assessment and exercise prescription. The investigators' intent is to pilot the program using a sample of patients. The objective of this pilot project:

To examine the effects of the late phase education session and home-based exercise program in restoring hip muscle strength, gait and function

ELIGIBILITY:
Inclusion Criteria:

* unilateral primary total hip arthroplasty (THA)
* 8-12 weeks post THA
* over the age of 18
* able to walk 15m without a walking aid
* able to participate in an exercise program without physical assistance
* available for follow up as per the study protocol
* able to read and understand English and follow verbal and visual instructions

Exclusion Criteria:

* medically unstable
* have central or peripheral nervous system deficits
* have an underlying terminal disease (cancer)
* have suspicion of infection following joint replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: orthopedic clinic outpatients (of one clinic)
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2009-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
hip muscle strength | 8-12 weeks post THA, 6-7 months post THA

SECONDARY OUTCOMES:
Gait | 8-12 weeks post THA, 6-7 months post THA

CONTACTS AND LOCATIONS:
Overall Officials: Ann Read, BScPT, MSc, Principal Investigator — CDHA
Locations (1):
- Orthopedic Clinic, QEII Health Sciences Centre, CDHA, Halifax, Nova Scotia, Canada